CLINICAL TRIAL: NCT03973463
Title: Effects of Diet Control and Resistance Exercise Training on Obesity Adults With Knee Osteoarthritis in Pain Relief, Body Composition, Lower Limb Function and Quality of Life
Brief Title: Effects of Diet Control and Resistance Exercise Training on Obesity Adults With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, yenyen0411, Dietitian，Investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201800607B0
Record Dates: First submitted 2019-05-30; First posted 2019-06-04 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Osteoarthritis, Knee; Obesity; Diet, Healthy; Training Group, Sensitivity
MeSH Terms: conditions — Osteoarthritis, Knee; Obesity; Hypersensitivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low fat diet,12 weeks low oil balance 1200 kcal / day (Sham Comparator): 12 weeks low oil balance 1200 kcal / day
  Interventions: Behavioral: Elastic knee joint movement
- 12-week resistance exercise 3 times a week (Experimental): 12-week stretch with resistance exercise, 3 times a week
  Interventions: Behavioral: Elastic knee joint movement
- 12 weeks low oil balance and resistance exercise (Experimental): 12 weeks low oil balance 1200 kcal / day and 12-week stretch with resistance exercise, 3 times a week
  Interventions: Behavioral: Elastic knee joint movement

INTERVENTIONS:
Behavioral: Elastic knee joint movement — Low resistance (7kg and 10kg) elastic band exercise 3 times a week for 12 weeks.Balanced diet reduces oil intake by 1200 calories per day. Maintains 12 weeks.Balanced diet reduces oil intake by 1200 calories per day. Maintains 12 weeks.
  Other Names: Low oil balanced diet 1200 kcal / day

SUMMARY:
The purpose of this study was to investigate the effects of obesity on knee degenerative arthritis on body composition after dietary control and elastic resistance exercise; and whether persistent exercise habits and dietary control can relieve pain and strengthen muscle strength. Improve the quality of life and the decline of other risk factors.

DETAILED DESCRIPTION:
Due to dietary westernization and overweight, the number of knee joint degeneration is increasing year by year. Degeneration of knee arthritis can lead to pain and not exercise, and thus other chronic diseases. When the weight loss exceeds 5.1%, the function of the knee joint can be significantly improved and low heat weight loss (1200 kcal / day) and very low heat weight loss (less than 800 kcal / day) both weight loss The results are equally good .Many studies have shown that early and mid-interventional resistance exercise can improve muscle weakness, pain and stiffness in patients with degenerative knee arthritis, and elastic resistance exercise can effectively improve lower limb function and increase physical activity in patients with knee arthritis However, there has been no research on the effects of diet control and resistance exercise training on pain relief, body composition, lower limb function and quality of life in obese knee degenerative arthritis. The purpose of this study was to explore the degenerative knee degeneration. The effect of arthritis on the composition of the body after a balanced diet calorie control and home-based low-intensity elastic resistance movement; and whether persistent exercise habits and diet control can relieve pain, strengthen muscle strength, improve quality of life and other risks The effect of factor decline. Expected to combine the diet control and home group exercise to improve the quality of life of patients with degenerative knee arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Cases of knee joint degeneration diagnosed by orthopedics, rheumatology and immunology physicians.
* X-ray interpretation (kellgren & Lawrence grade) grades 1 to 3 or mild to moderate patients.
* Willing to sign written consent form.
* Pain Index (VAS) ≧ 4/10.
* Men and women over the age of 55.
* Body mass index (BMI) ≧ 27 kg/m^2.

Exclusion Criteria:

* Unable to act on your own.
* X-ray interpretation (kellgren & Lawrence level) is greater than level 3 or is a serious level.
* Patients who have undergone knee arthroplasty on one or both feet.
* Patients with terminal liver and kidney disease.
* Those who are unable to perform physical function measurement after severe diagnosis of heart and lung disease after diagnosis by the physician.
* High blood pressure with poor control (systolic blood pressure greater than or equal to 180 mmHg at the time of return).
* Pregnant women or breastfeeding women.
* Those who have coronary stents, cardiac rhythms, or other metallic substances in the body are not recommended for total body composition analysis.
* Those with severe hip, knee, and lower back pain who are unable to perform exercise, other neuromuscular, skeletal joints, or rheumatic diseases may be exacerbated by exercise. Or those who have musculoskeletal injuries in the past six months (such as bruises, fractures, etc.).
* Unable to cooperate with the test or halfway through the test.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-05-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
WOMAC | Baseline and after 3 months
  WOMAC is used to measure the patient's home knee function. Each question is scored using a five-point scale. The higher the score, the worse the knee function.
  This study assessed the amount of change in WOMAC scores, whether it was lower than baseline after 12 weeks.
KOOS | Baseline and after 3 months
  KOOS is based on WOMAC and covers a wider range. The score of each topic is 0-4 points. The higher the score after the conversion formula, the better the knee joint function. This study assessed changes in KOOS scores, whether it was higher than baseline after 12 weeks.
Body fat percentage | Baseline and after 3 months
  Assess the amount of body fat (%) change, whether it can be less than baseline after 12 weeks
Body Mass Index | Baseline and after 3 months
  Assess the amount of Body Mass Index(kg/m^2) change, whether it can be less than baseline after 12 weeks
waistline | Baseline and after 3 months
  Waist circumference change from baseline to 12 weeks (cm)

SECONDARY OUTCOMES:
hand grip force measurement | Baseline and 3 months
  Easy to stand. Used to grasp the grip
2.44m time up to go | Baseline and 3 months
  Stand up when you hear the start password. Use the brisk walk to bypass the marker point and then return to the chair to sit down.
30 chair stand test | Baseline and 3 months
  Sit down and stand up to stand upright, then quickly return to sit down for an action, within 30 seconds
total cholesterol | Baseline and 3 months
  Cases will be tested for total cholesterol (mg/dL) in routine outpatient care. This study, at baseline and 12 weeks later, copied the most recent total cholesterol report from the case.
  The amount of change in total cholesterol after baseline and 12 weeks was compared.
Low-density cholesterol | Baseline and 3 months
  Cases in the outpatient routine care will be blood tests for low-density cholesterol (LDL-C, mg / dL), the study of the most recent low-density cholesterol report from the case at baseline and 12 weeks later, compared with baseline and 12 weeks later Low-density cholesterol has changed.
triglyceride | Baseline and 3 months
  Cases will be tested for triglycerides (mg/dL) in routine outpatient care. In the study, at the baseline and after 12 weeks, the most recent triglyceride report from the case was copied.
  The amount of change in triglyceride at baseline and after 12 weeks was compared.

CONTACTS AND LOCATIONS:
Overall Officials: YEN-I HSU, Study Director — Chang Gung Medical Foundation
Locations (1):
- Chang Gung Medical Foundation, Taipei, Taiwan, Republic of China, Taiwan